CLINICAL TRIAL: NCT05600348
Title: Personalized Pork: Dose-dependent Identification of Unique Biomarkers
Brief Title: Dose-dependent Identification of Unique Biomarkers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Responsible Party: Principal Investigator, Shirin Hooshmand, Professor, San Diego State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: 5A949A
Record Dates: First submitted 2022-10-22; First posted 2022-10-31 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2023-12

CONDITIONS: Healthy
Keywords: Metabolome; Pork; Metabolite

STUDY DESIGN:
Intervention Model Description: 3 conditions, order randomly allocated
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 0 oz Pork (Experimental): Participants receive 0 oz pork and 6 oz 50:50 blend of chicken and beef per day
  Interventions: Dietary Supplement: Pork Consumption
- 3 oz Pork (Experimental): Participants receive 3 oz pork and 3 oz 50:50 blend of chicken and beef per day
  Interventions: Dietary Supplement: Pork Consumption
- 6 oz Pork (Experimental): Participants receive 6 oz pork and 0 oz 50:50 blend of chicken and beef per day
  Interventions: Dietary Supplement: Pork Consumption

INTERVENTIONS:
Dietary Supplement: Pork Consumption — Feeding of pork is controlled at 0, 3 or 6 oz per day for 4 weeks each in random order.

SUMMARY:
The purpose of the research is to assess the dose-dependent impacts of the consumption of fresh pork on blood-borne metabolites (markers) following the controlled feeding of pork

DETAILED DESCRIPTION:
Eligible participants will follow 3 randomly ordered 4-week feeding periods varying only with the consumption of 0, 3 or 6 oz of pork or a 50:50 blend of chicken and beef (6, 3 and 0 oz for respective trials to ensure similar total poultry/meat intake among trials).

ELIGIBILITY:
Inclusion Criteria:

* generally healthy (i.e., an absence of diagnosed chronic illnesses and inborn metabolic disorders)
* Age 18-65
* all races
* both sexes
* willingness to comply with the research diet requirements

Exclusion Criteria:

* special dietary needs (e.g., vegetarianism, gluten-free, etc.)
* use of medication known to influence metabolism
* smoking
* substance use

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Metabolic biomarker discovery | 4 weeks
  Biomolecules detected through metabolomic profiling that will result in discovery of a metabolic signature for pork intake

SECONDARY OUTCOMES:
Fasted Glucose | 4 weeks
  Fasted Glucose
Insulin | 4 weeks
  Insulin
HDL Cholesterol | 4 weeks
  HDL Cholesterol
Total Cholesterol | 4 weeks
  Total Cholesterol
LDL-Cholesterol | 4 weeks
  LDL-Cholesterol
Triglycerides | 4 weeks
  Triglycerides
Interleukin-6 | 4 weeks
  Interleukin-6
C-Reactive Protein | 4 weeks
  C-Reactive Protein
Blood Pressure | 4 weeks
  Systolic and Diastolic
Body Composition | 4 weeks
  Weight measured via scalre, body fat% muscle mass as measured via DEXA

CONTACTS AND LOCATIONS:
Overall Officials: Shirin Hooshmand, PhD, Principal Investigator — San Diego State University
Locations (1):
- School of Exercise and Nutritional Sciences, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No